CLINICAL TRIAL: NCT01948232
Title: A Phase II Open Label Pilot Study of the Angiotensin-converting Enzyme Inhibitor, Perindopril, in Pediatric Cancer Survivors With Evidence of Early Cardiac Remodelling or Dysfunction.
Brief Title: Pilot Study of Perindopril in Childhood Cancer Survivors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Paul Nathan, Director, AfterCare Program; Staff Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000035483
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Childhood Cancer Survivors
MeSH Terms: interventions — Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perindopril (Experimental)
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Perindopril — Angiotensin converting enzyme inhibitor
  Other Names: Coversyl

SUMMARY:
The purpose of this study is to evaluate the feasibility of conducting a medical intervention trial in childhood cancer survivors with early echocardiographic evidence of cardiac remodeling.

DETAILED DESCRIPTION:
Anthracycline cardiotoxicity is characterized by ventricular remodeling and progressive cardiac dysfunction. Since ventricular remodeling in other types of heart failure can be treated effectively with an angiotensin-converting enzyme inhibitor (ACEi), these agents would appear a logical therapy in children with anthracycline-induced heart failure. Previous experience with ACEi in childhood cancer survivors has shown mixed results, possibly due to the fact that treatment is initiated too late in the natural history of the disease. Providing treatment in childhood cancer survivors with early signs of cardiac remodeling may be more effective than treating children who have global dysfunction. The benefits of early intervention are unclear, so it is unclear whether CCS and their parents will be willing to receive treatment where the target outcome (prevention of decreased global function or congestive heart failure) may not occur for years after the intervention. Assessing the feasibility of this pre-emptive approach is the primary aim of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the Survivor Cohort of the PCS2 study at The Hospital for Sick Children at the time of enrollment.
2. Aged < 20 years at enrollment.
3. Weight ≥ 25kg at enrollment
4. LVPW Z-score ≤-2.0 at any of the 0, 12 or 24 month PCS2 echocardiography assessments, on two consecutive echocardiograms at least 3 but no more than 15 months apart.
5. EF greater than 50% at enrollment
6. Serum potassium (to be ˃5.0mMol/l) at Initiation

Exclusion Criteria:

1. Known associated cardiac conditions for which angiotensin converting enzyme therapy is contraindicated (such as aortic stenosis, severe coarctation of the aorta, or hypertrophic cardiomyopathy with LV outflow tract obstruction)
2. Active malignancy detected within last 2 years (i.e. must be at least 2 years in remission)
3. Prior radiation therapy to a field that involved the heart
4. Prior symptomatic heart failure, or prior reduction in EF below 50% detected on surveillance echocardiography.
5. Use of any cardioactive medications including diuretics within the last 6 months
6. Concurrent serious or life threatening disease or extracardiac organ compromise which would limit participation in the trial or potentially have secondary effects on cardiac function, as determined by the treating physician.
7. Renal dysfunction precluding ACEi therapy, defined as serum creatinine greater than the 95th percentile for age or eGFR by the modified Schwartz formula of less than the 5th percentile prior to recruitment to the interventional trial (within 30 days of recruitment date)
8. Hypertension requiring treatment.
9. History of angioedema or ACEi hypersensitivity
10. Patients with hereditary problems of galactose intolerance, glucose-galactose malabsorption, or the Lapp lactase deficiency.
11. Upper airway obstructive lesions
12. Pregnancy
13. Breast-feeding

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients consenting to study | 18-month
  The number of eligible patients approached to join the study, the proportion consenting to the study, the proportion refusing the study (with reasons for refusal) and the proportion remaining on study at 18-months.

SECONDARY OUTCOMES:
LV wall thinning | 18 months
  Rate of change of the end-diastolic left ventricular posterior wall z-score and of the thickness to dimension ratio z-score

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada